CLINICAL TRIAL: NCT05526105
Title: Gastric Ultrasound in Critically Ill Patients for Evaluation of Gastric Volume Residuals; A Comparison of NPO Protocols
Brief Title: Gastric US in ICU Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Laura M. Chiang, Assistant Professor of Anesthesiology at the Geisel School of Medicine, Co-medical Director of the Surgical Intensive Care Unit, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY02001249
Record Dates: First submitted 2022-08-15; First posted 2022-09-02 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Surgery; Aspiration Pneumonia
Keywords: NPO Protocols; Intensive Care Unit; Gastric Ultrasound; Ultrasound; Surgical Intensive Care Unit; NPO; Nasogastric Tube; Orogastric Tube; Enteral Nutrition; Parenteral Nutrition; Gastric Residual Volume; Aspiration; Critical Illness Nutrition
MeSH Terms: conditions — Critical Illness; Pneumonia, Aspiration; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to be NPO after midnight (standard protocol) or feed up until call to OR then decompressed (liberal protocol).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard ASA NPO Protocol (Experimental): Patients will be made NPO at midnight prior to date of surgery.
  Interventions: Diagnostic Test: Gastric Ultrasound
- Liberal Feeding Protocol (Experimental): Patients will be fed enterally up until call to OR at which time their stomachs will be decompressed with a pre-existing gastric tube.
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — Gastric ultrasound in the supine and right lateral decubitus position for patients going for operative intervention with a protected airway.

SUMMARY:
This is a case series study using gastric ultrasound in critically ill patients to quantify gastric residual volumes to compare the efficacy of different NPO protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older, admitted to the ICU, requiring general anesthesia or sedation for a procedure with a pre-existing, cuffed endotracheal or tracheostomy tube. Most patients admitted to the ICU would be unable to consent.

Exclusion Criteria:

* Known upper gastrointestinal anatomical problem that would prevent accurate estimation of gastric volume, gastric perforation, pregnancy beyond the first trimester.
* Lack of a pre-existing, cuffed endotracheal or tracheostomy tube.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-02-03 (Estimated); Study Completion 2025-02-03 (Estimated)

PRIMARY OUTCOMES:
Gastric Residual Volumes | Within one hour of operative intervention.
  Quantification of gastric residual volumes as measured in milliliters using antral cross-sectional areas and semi-quantitative gastric volumes using standardized grading scores.

SECONDARY OUTCOMES:
Comparison of two different NPO protocol populations | Within four months of study completion, 16 months from study start
  Comparing standard ASA NPO protocol vs liberal, feed-up-until-call to OR protocol as defined by comparison of gastric volumes (mLs).
Peri-operative aspiration events | Within four months of study completion, 16 months from study start
  Number of aspiration events per number of operative interventions.
Estimation of the amount of enteral nutrition lost prior to surgery using the different NPO protocols | Zero to sixteen hours prior to surgery
  Calculation of enteral nutrition held during NPO time in kilocalories.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Chiang, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No